CLINICAL TRIAL: NCT02531360
Title: Phase 0 Evaluation of [18F]MNI-815 as a Potential PET Radioligand for Imaging Tau Protein in the Brain of Patients With Alzheimer's Disease and Other Tauopathies
Brief Title: Evaluation of [18F]MNI-815 as a Potential PET Radioligand for Imaging Tau Protein in the Brain of Patients With Tauopathies
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Molecular NeuroImaging (Other)
Collaborators: Life Molecular Imaging SA (Industry)
Responsible Party: Principal Investigator, Danna Jennings, Principal Investigator, Molecular NeuroImaging
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MNI-815
Record Dates: First submitted 2015-06-09; First posted 2015-08-24 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease (AD); Progressive Supranuclear Palsy (PSP); Cortical Basal Syndrome (CBS); Frontal Temporal Dementia (FTD)
MeSH Terms: conditions — Alzheimer Disease; Supranuclear Palsy, Progressive | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]MNI-815 (MNI-815) (Experimental): At the [18F]MNI-815 PET imaging visit, subjects will be injected with no more than 10mCi of [18F]MNI-815
  Interventions: Drug: [18F]MNI-815 (MNI-815)

INTERVENTIONS:
Drug: [18F]MNI-815 (MNI-815) — All enrolled subjects will undergo an [18F]MNI-815 PET imaging visit. As a part of the screening visit, subjects will undergo [18F]florbetaben (FBB) PET imaging to determine if they have significant amyloid deposition.
  Other Names: [18F]MNI-815; FBB; [18F]Florbetaben

SUMMARY:
The overall goal of this imaging trial is to characterize [18F]MNI-815, a PET radioligand for imaging Tau.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are child-bearing potential, must commit to use of a barrier contraception method for the duration of the study.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration
* Willing and able to cooperate with study procedures

Healthy Control subjects:

* Males and females aged between 50 - 70 years. Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the [18F]MNI-815 imaging visit.
* No cognitive impairment from neuropsychological battery as judged by the investigator
* Have a CDR score=0
* Has FBB PET imaging demonstrating no evidence for significant amyloid binding based on qualitative (visual read) and quantitative analysis.
* Modified Hachinski Ischemia Scale score of ≤ 4.

Prodromal or Moderate Alzheimer's Disease subjects:

* Males and females aged between 50 - 90 years.
* Have prodromal or moderate Alzheimer's disease, based on the NINCDS/ADRDA and DSM-IV criteria.
* Have a CDR score of 0.5 for prodromal AD subjects and CDR > 1.0 for moderate AD subject at screening.
* Has a FBB PET imaging demonstrating amyloid binding based on qualitative (visual read) and quantitative analysis.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* A brain MRI that supports a diagnosis of AD, with no evidence of focal disease to account for dementia or MRI exclusion criteria.
* Medications taken for symptomatic treatment of AD must be maintained on a stable dosage regimen for at least 1 month before the [18F]MNI-815 imaging visit.
* The subject has an appropriate caregiver capable of accompanying subject on all visits.
* Signed and dated written informed consent obtained from the subject and, when applicable, the subject's legally authorized representative or caregiver.

Frontotemporal Dementia subjects:

* Has a clinical diagnosis of FTD based on consensus for clinical diagnosis of frontotemporal dementia criteria (Neary, et al 1998)
* Has a FBB PET imaging demonstrating no evidence of significant amyloid binding based on qualitative (visual read) and quantitative analysis.
* A brain MRI that supports a diagnosis of FTD, with no evidence of focal disease to account for dementia or MRI exclusion criteria.
* Medications taken for symptomatic treatment of cognitive dysfunction must be maintained on a stable dosage regimen for at least 1 month before the screening visit.
* The subject has an appropriate caregiver capable of accompanying subject on all visits to the center.
* Signed and dated written informed consent obtained from the subject and, when applicable, the subject's legally authorized representative or caregiver.
* Modified Hachinski Ischemia Scale score of ≤ 4.

Progressive Supranuclear Palsy subjects:

* Has a clinical diagnosis of PSP based the NINDS and Society for PSP criteria (Litvan, et al 1996)
* Has FBB PET imaging demonstrating no evidence of significant amyloid binding based on qualitative (visual read) and quantitative analysis.
* A brain MRI that supports a diagnosis of PSP, with no evidence of focal disease to account for dementia or MRI exclusion criteria.
* Medications taken for treatment of PSP symptoms must be maintained on a stable dosage regimen for at least 1 month before the screening visit.
* The subject has an appropriate caregiver capable of accompanying subject on all visits to the center.
* Signed and dated written informed consent obtained from the subject and, when applicable the subject's legally authorized representative or caregiver.
* Modified Hachinski Ischemia Scale score of ≤ 4.

Corticobasal Syndrome Subjects:

* Has a clinical diagnosis of CBS based on consensus criteria for possible or probable corticobasal degeneration (Armstrong et al, 2013)
* Has a FBB PET imaging demonstrating no evidence of significant amyloid binding based on qualitative (visual read) and quantitative analysis.
* A brain MRI that supports a diagnosis of CBS, with no evidence of focal disease to account for dementia or MRI exclusion criteria.
* Medications taken for treatment of CBS symptoms must be maintained on a stable dosage regimen for at least 1 month before the screening visit.
* The subject has an appropriate caregiver capable of accompanying subject on all visits to the center.
* Signed and dated written informed consent obtained from the subject and, when applicable, the subject's legally authorized representative or caregiver.
* Modified Hachinski Ischemia Scale score of ≤ 4.

Exclusion Criteria:

For all subjects

* Current or prior history of any alcohol or drug abuse.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure is >15 mSv and would exceed the annual limits.
* Pregnancy or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* MRI exclusion criteria include: Pathology that may be responsible for the neurologic status of the patient such as infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with CNS disease,
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.

Exclusion criteria for subjects with AD subjects:

* Has received treatment that targeted amyloid-beta or tau within the last 24 months.
* Has a FBB PET imaging demonstrating no evidence of significant amyloid binding irrespective of other previous measurements of beta amyloid that may be available for review.

Exclusion criteria for subjects with PSP or CBS subjects:

* Has FBB PET imaging with evidence of significant amyloid binding irrespective of other previous measurements of beta amyloid that may be available for review.
* Has received treatment that targeted tau within the last 24 months.
* Have any other neurological condition other than CBS or PSP that could account for cognitive or motor deficits including: Specifically:
* A diagnosis of idiopathic Parkinson's disease or Lewy body dementia and/or have a prominent and sustained response to levodopa therapy;
* History of repeated strokes with stepwise progression of parkinsonian features or history of major stroke

FTD subjects:

* Has FBB PET imaging with evidence of significant amyloid binding irrespective of other previous measurements of beta amyloid that may be available for review.
* Has received treatment that targeted tau within the last 24 months.

Healthy subjects:

•Has FBB PET imaging with evidence of significant amyloid binding irrespective of other previous measurements of beta amyloid that may be available for review.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Brain uptake of [18F]MNI-815 | 18 months
  The PET imaging outcome measure to evaluate tau burden will be the standardized uptake value (SUV), which will be calculated for the areas of interest by using the established methods for normalizing to subject weight and injected dose.

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Molecular NeuroImaging, LLC
Locations (1):
- Molecular NeuroImaging, LLC, New Haven, Connecticut, United States

REFERENCES:
- [Background] Neary D, Snowden JS, Gustafson L, Passant U, Stuss D, Black S, Freedman M, Kertesz A, Robert PH, Albert M, Boone K, Miller BL, Cummings J, Benson DF. Frontotemporal lobar degeneration: a consensus on clinical diagnostic criteria. Neurology. 1998 Dec;51(6):1546-54. doi: 10.1212/wnl.51.6.1546. PMID 9855500
- [Background] Litvan I, Agid Y, Calne D, Campbell G, Dubois B, Duvoisin RC, Goetz CG, Golbe LI, Grafman J, Growdon JH, Hallett M, Jankovic J, Quinn NP, Tolosa E, Zee DS. Clinical research criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome): report of the NINDS-SPSP international workshop. Neurology. 1996 Jul;47(1):1-9. doi: 10.1212/wnl.47.1.1. PMID 8710059
- [Background] Armstrong MJ, Litvan I, Lang AE, Bak TH, Bhatia KP, Borroni B, Boxer AL, Dickson DW, Grossman M, Hallett M, Josephs KA, Kertesz A, Lee SE, Miller BL, Reich SG, Riley DE, Tolosa E, Troster AI, Vidailhet M, Weiner WJ. Criteria for the diagnosis of corticobasal degeneration. Neurology. 2013 Jan 29;80(5):496-503. doi: 10.1212/WNL.0b013e31827f0fd1. PMID 23359374
- See also: Molecular NeuroImaging — http://www.mnimaging.com
- See also: Institute for Neurodegenerative Disorders — http://indd.org